CLINICAL TRIAL: NCT03355248
Title: The Effect of Decreased Opioid Prescribing on Pain Control and Patient Satisfaction Following Cesarean Section
Brief Title: Satisfaction Following Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ProMedica Health System (Other)
Responsible Party: Principal Investigator, James Van Hook, Medical Doctor, ProMedica Health System
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB #17-064
Record Dates: First submitted 2017-11-17; First posted 2017-11-28 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Pain, Postoperative; Cesarean Section Complications; Postpartum Disorder; Opioid Use
Keywords: postpartum; postoperative cesarean pain management; opioid requirements
MeSH Terms: conditions — Pain, Postoperative; Puerperal Disorders | interventions — oxycodone-acetaminophen

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants are blinded to the group assignment and are not made aware of what interventions are being assigned, only that pain management and satisfaction are being evaluated
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group - 28 (Active Comparator): The control group (post-operative cesarean section) will be prescribed 28 Oxycodone Acetaminophen at the time of discharge. Both groups will also be provided with a handout on non-opioid analgesia. The groups will be assigned randomly in blocks. Specifically, the first half of the patients will automatically be placed in the experimental arm and the second half into the control arm of the study
  Interventions: Other: Oxycodone Acetaminophen
- Experimental - 20 (Experimental): The experimental group (post-operative cesarean section) will be prescribed 20 Oxycodone Acetaminophen at the time of discharge. Both groups will also be provided with a handout on non-opioid analgesia. The groups will be assigned randomly in blocks. Specifically, the first half of the patients will automatically be placed in the experimental arm and the second half into the control arm of the study
  Interventions: Other: Oxycodone Acetaminophen

INTERVENTIONS:
Other: Oxycodone Acetaminophen — Decrease in opioid prescribing for post-operative cesarean pain management
  Other Names: Percocet

SUMMARY:
Presently, the standard of care at the investigators' practice is that the discharging physician decides the type and amount of opioid medication to prescribe a patient following a cesarean section. After informed consent has been obtained, patients will be enrolled in this randomized-controlled equivalence study. The experimental group will be prescribed 20 oxycodone-acetaminophen and the control group will be prescribed 28 oxycodone-acetaminophen at the time of discharge. Both groups will also be provided with a handout on non-opioid analgesia. The groups will be assigned randomly in blocks. The investigators will recruit patients either in the clinic, if participants are to have a scheduled cesarean section, or at some time during the hospital admission for delivery. The satisfaction survey and pain scale will be administered at the postoperative check by the clinic staff and providers. These surveys will be stored in a secure location at the clinic. If the patient does not show up for their postoperative visit, 3 attempts total will be made by an investigator to reach the patient and administer both surveys by phone within 2 weeks of discharge. A preliminary analysis of the data will be done once half the study patients have been recruited. The investigators do not foresee any threats to the external or internal validity of the study. The investigators are taking many measures to limit study bias. First, block randomization will help limit discrepancies between groups. Also, strict adherence to the inclusion and exclusion criteria will also help limit confounders that may make data difficult to interpret, such as non-opioid naïve patients and complications that may potentially increase pain and opioid requirements. Lastly, blinding of patients to the number of pills participants receive will help mitigate patient bias.

DETAILED DESCRIPTION:
Presently, the standard of care at our practice is that the discharging physician decides the type and amount of opioid medication to prescribe a patient following a cesarean section. After informed consent has been obtained, patients will be enrolled in our randomized-control, equivalence study. The experimental group will be prescribed 20 oxycodone-acetaminophen and the control group will be prescribed 28 oxycodone-acetaminophen at the time of discharge. Both groups will also be provided with a handout on non-opioid analgesia. The groups will be assigned randomly in blocks. The investigators will recruit patients either in the clinic, if participants are to have a scheduled cesarean section, or at some time during the hospital admission for delivery. The satisfaction survey and pain scale will be administered at the postoperative check by the clinic staff and providers. If the patient does not show up for their postoperative visit, 3 attempts total will be made by an investigator to reach the patient and administer both surveys by phone within 2 weeks of discharge. A preliminary analysis of the data will be done once half the study patients have been recruited. First, block randomization will help limit discrepancies between groups.

Subject evaluation will generally be limited to no more than 3 weeks following surgery. Evaluations will occur at the postoperative visit via two surveys (see below). If the patient does not show up for the clinic visit, 3 attempts will be made by an investigator to reach the patient and administer both surveys by phone within 2 weeks of discharge.

Variables of interest:

1. Age
2. Race
3. Insurance
4. Repeat cesarean section
5. Classification of cesarean section (scheduled, unscheduled, emergent)
6. Type of skin incision and closure
7. Urine toxicology screen results
8. Tubal ligation at the time of cesarean
9. Anesthesia (General or regional [epidural, spinal or combined], if regional, duramorph given)
10. Length of hospital stay
11. Number of refills

ELIGIBILITY:
Inclusion Criteria:

1. Center for health services (CHS) patient
2. Cesarean section
3. >/= 18 years of age

Exclusion Criteria:

1. Non-CHS patients (i.e. regional or private)
2. <18 years of age
3. Allergy to hydrocodone, oxycodone, acetaminophen or NSAIDs
4. Contraindication to using medications (i.e hypertensive disorders of pregnancy)
5. Hospitalization >7 days, which suggest complications that may increase pain and opioid requirements
6. Complications (wound infections, re-explorations, cesarean hysterectomies, etc…)
7. Urine toxicology screen positive for opioids on admission
8. Recent use as defined by either patient reported use of opioids within the last 30 days or an Ohio Automated Rx Reporting System (OARRS) reports that shows prescription of opioids within 30 days of admission for delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Postpartum cesarean patients
Enrollment: 60 (Actual)
Dates: Start 2017-08-18 (Actual); Primary Completion 2020-08-14 (Actual); Study Completion 2020-08-14 (Actual)

PRIMARY OUTCOMES:
Post-cesarean pain management | 1 week post-op cesarean
  Our main aim is to determine the effect of decreased opioid prescribing on pain control following cesarean section. Our hypothesis is that despite decreased opioid prescribing [20 oxycodone-acetaminophen (5/325mg)] following cesarean section, pain scores will be equivalent to the control group [28 oxycodone-acetaminophen (5/325mg)]. Pain control will be measured by an 11-point numeric scale.

SECONDARY OUTCOMES:
Post-cesarean patient satisfaction with management | 1 week post-op cesarean
  Secondary outcomes include patient satisfaction as assessed by a survey

CONTACTS AND LOCATIONS:
Overall Officials: James Van Hook, MD, Principal Investigator — ProMedica Health System
Locations (1):
- Center for Health Services, Toledo, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Centers for Disease Control and Prevention. Wide-ranging Online Data for Epidemiologic Research (WONDER), Multiple-Cause-of-Death file, 2000-2014. 2015. Available at: http://www.cdc.gov/nchs/data/health_ policy/AADR_drug_poisoning_involving_OA_Heroin_US_2000-2014.pdf. Accessed June 9, 2017.
- [Background] Rudd RA, Seth P, David F, Scholl L. Increases in Drug and Opioid-Involved Overdose Deaths - United States, 2010-2015. MMWR Morb Mortal Wkly Rep. 2016 Dec 30;65(50-51):1445-1452. doi: 10.15585/mmwr.mm655051e1. PMID 28033313
- [Background] Hill MV, Stucke RS, McMahon ML, Beeman JL, Barth RJ Jr. An Educational Intervention Decreases Opioid Prescribing After General Surgical Operations. Ann Surg. 2018 Mar;267(3):468-472. doi: 10.1097/SLA.0000000000002198. PMID 28267689
- [Background] Bartels K, Mayes LM, Dingmann C, Bullard KJ, Hopfer CJ, Binswanger IA. Opioid Use and Storage Patterns by Patients after Hospital Discharge following Surgery. PLoS One. 2016 Jan 29;11(1):e0147972. doi: 10.1371/journal.pone.0147972. eCollection 2016. PMID 26824844
- [Background] Hill MV, McMahon ML, Stucke RS, Barth RJ Jr. Wide Variation and Excessive Dosage of Opioid Prescriptions for Common General Surgical Procedures. Ann Surg. 2017 Apr;265(4):709-714. doi: 10.1097/SLA.0000000000001993. PMID 27631771
- [Background] Bateman BT, Cole NM, Maeda A, Burns SM, Houle TT, Huybrechts KF, Clancy CR, Hopp SB, Ecker JL, Ende H, Grewe K, Raposo Corradini B, Schoenfeld RE, Sankar K, Day LJ, Harris L, Booth JL, Flood P, Bauer ME, Tsen LC, Landau R, Leffert LR. Patterns of Opioid Prescription and Use After Cesarean Delivery. Obstet Gynecol. 2017 Jul;130(1):29-35. doi: 10.1097/AOG.0000000000002093. PMID 28594763
- [Background] Osmundson SS, Schornack LA, Grasch JL, Zuckerwise LC, Young JL, Richardson MG. Postdischarge Opioid Use After Cesarean Delivery. Obstet Gynecol. 2017 Jul;130(1):36-41. doi: 10.1097/AOG.0000000000002095. PMID 28594766
- [Background] Prabhu M, McQuaid-Hanson E, Hopp S, Burns SM, Leffert LR, Landau R, Lauffenburger JC, Choudhry NK, Kaimal A, Bateman BT. A Shared Decision-Making Intervention to Guide Opioid Prescribing After Cesarean Delivery. Obstet Gynecol. 2017 Jul;130(1):42-46. doi: 10.1097/AOG.0000000000002094. PMID 28594762
- [Background] Manchikanti L, Helm S 2nd, Fellows B, Janata JW, Pampati V, Grider JS, Boswell MV. Opioid epidemic in the United States. Pain Physician. 2012 Jul;15(3 Suppl):ES9-38. PMID 22786464